CLINICAL TRIAL: NCT01422668
Title: Effect of Coffee Consumption on the Glycemic Index of Khalas Dates Tested in Healthy and Diabetic Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: United Arab Emirates University (Other)
Responsible Party: Principal Investigator, Juma Alkaabi, Assistant Professor of Medicine, Faculty of Medicine and Health Sciences, United Arab Emirates University
Allocation: Non-Randomized | Model: Single Group | Masking: Single
Other Study IDs: UAEU: GI Dates Study
Record Dates: First submitted 2011-08-18; First posted 2011-08-24 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Diabetes Mellitus
Keywords: Glycemic index; Dates; Diabetes; Coffee
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GI of Khalas dates (Active Comparator): The Glycemic indices of the Khalas dates were measured for healthy and diabetic subjects.
  Interventions: Other: Khalas dates
- GI of the Khalas dates with Coffee (Experimental): measuring the effect of 100 ml of coffee consumption on the GI of the Khalas dates among healthy and diabetic subjects.
  Interventions: Other: Khalas dates

INTERVENTIONS:
Other: Khalas dates — every subject recieved 50 grams reducing carbohydrates equivalent of khalas dates

SUMMARY:
The aim of this study was to evaluate the composition of Khalas, a very common type of dates used in the UAE and to determine the effects of drinking Arabic coffee on the results of GI tests in both healthy and diabetic subjects.

DETAILED DESCRIPTION:
Background:The consumption of dates along with coffee is a deeply rooted habit in many societies. This study was designed to determine the effect of coffee consumption on the glycemic index of a common variety of dates (Khalas) tested in healthy subjects and individuals with type 2 diabetes mellitus.

Methods:Composition analysis was carried out for Khalas dates (Tamer stage) and the weight of the dates flesh equivalent to 50 g of available carbohydrate was calculated. The study subjects were thirteen healthy volunteers with a mean (± SD) age of 40.2 ± 6.7 years and ten participants with type 2 diabetes mellitus (controlled on lifestyle measures and/or metformin) with a mean HbA1c (± SD) of 6.6 ± (0.7 %) and a mean age (± SD) of 40.8 ± 5.7 years. Each subject was tested on five separate days with 50 g of glucose (on 3 occasions) and 50 g equivalent of available carbohydrates from the dates without coffee (on one occasion) and with coffee (on another occasion). Capillary glucose was measured in the healthy subjects at 0, 15, 30, 45, 60, 90 and 120 min and for the diabetics at 0, 30, 60, 90, 120, 150 and 180 min. The glycemic indices were determined as ratios of the incremental areas under the response curves for the dates alone/with coffee compared to glucose. Statistical analyses were performed using Student's t-tests.

ELIGIBILITY:
Inclusion Criteria:

* required that those in the healthy group were healthy and in the diabetes group that their diabetes was controlled (HbA1c ≤8%) on diet with or without metformin

Exclusion Criteria:

* morbid obesity (BMI > 40 kg/m2)
* pre diabetes
* pregnancy
* presence of gastroenterological disorders
* alimentary tract surgery
* a history of gastroenteritis in the prior six months
* any alcohol intake
* smoking
* taking any medications (except metformin)
* poorly controlled diabetes (HbA1c > 8%) and the presence of acute or chronic diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Glycemic Index of Khalas dates with and without coffee | 2 or 3 hours
  Every subject recieved 50 grams reducing sugars of Khalas dates with and without coffee. Measuring glucose level over 2 hours in Healthy subjects and over 3 hours in diabetic subjects as per a standard protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Juma M Alkaabi, MD, Principal Investigator — Assistant professor Internal Medicine Department FMHS UAE University; Bayan Al-Dabbag, PhD, Study Chair — FMHS UAE university; Hussein Saadi, MD, Study Chair — Professor of Medicine, FMHS UAE University; Salah Gariballa, MD, Study Chair — Professor of Medicine FMHS UAE University; Yasin Javed, Msc, Study Chair — FMHS UAE University
Locations (1):
- Faculty of Medicine and Health Sciences UAE University, Al Ain City, AB, United Arab Emirates